CLINICAL TRIAL: NCT05304260
Title: Prevalence of Dental Anomalies in Deciduous Dentition and Risk Factors Associated With Non-syndromic Oral Clefts Patients: A Cross-sectional Study.
Brief Title: Prevalence of Dental Anomalies in Oral Clefts Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Saada Mohammed Ibrahim El-Aarag, Principal investigator, Cairo University
Other Study IDs: prevalence of dental anomalies
Record Dates: First submitted 2022-02-12; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Anomaly
Keywords: dental anomalies
MeSH Terms: conditions — Congenital Abnormalities; Tooth Abnormalities | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical and radiographic examination — Prevalence of dental anomalies in deciduous dentition and risk factors associated with non-syndromic oral clefts patients: A cross-sectional study.

SUMMARY:
To assess the prevalence of dental anomalies in the deciduous dentition in children with oral clefts and to investigate the associated risk factors.

DETAILED DESCRIPTION:
Oral clefts lip and/or palate are considered as the most common oro-facial defects in children with an unclear complex etiology.

The international prevalence in newborns was estimated as 14 per 10,000 live births worldwide. Around 70% of cases occur as a non-syndromic cleft lip and/or cleft palate (NSCL/P)], and the resting 30% are associated with Mendelian disorders or teratogenic, chromosomal and sporadic conditions.

Non syndromic cleft lip and/or palate divided into cleft lip (CL), cleft lip and palate (CL/P) and cleft palate (CP) based on epidemiological features and embryologic timing.

The exact etiology is not completely known, but attributed to a mixture of genetic and environmental factors. The usefulness of epidemiological knowledge is important in assessing the burden of oral clefts in order to plan public health resources. Also, knowing the causes of oral clefts, which stimulates research on primary prevention and treatments to improve the quality of health and care.

The incidence of dental defects in cleft patients can be used as clinical indicators for defining cleft sub-phenotypes, as well as providing numbers of instances.

Dental anomalies in children can lead to an increased risk of dental problems from esthetic to orthodontic problems. In Egypt, there is lacking of information on the occurrence of dental defects in the deciduous dentition of children with oral clefts. Also oral clefts are complicated epidemiological condition and further investigations are needed to know about the risk factors of this situation.

ELIGIBILITY:
Inclusion Criteria:

* Children with oral cleft lip and/or palate with ages varying from 4 to 6 years.
* Children with primary dentition.
* Parents who accept to participate in the study.
* Compliant children.

Exclusion Criteria:

* Healthy children and their guardians
* Syndromic oral clefts children

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: oral clefts children
Sampling Method: Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental anomalies | baseline
  measurement method: clinical and radiographic examination used to asses prevalence of dental anomalies, unit of measurement binary (yes, no).

SECONDARY OUTCOMES:
Predisposing risk factors for oral clefts | baseline
  Measurement method: questionnaire used to assess risk factors of oral clefts, measurement unit: binary questions (yes, no).

REFERENCES:
- [Background] 1. Carolina, A., Cordeiro, S., Isabel, ;, Olegário Da Costa, C., Carmela, ;, Bresolin, R., Carlos, J., & Imparato, P. (2018). Calidad de vida relacionada con la salud oral, características socioeconómicas y de comportamiento de los pacientes fisurados menores de 7 años Artículo Original (Vol. 8, Issue 1).
- [Background] Qi L, Liu J, Zhang Y, Wang J, Yang M, Gong T, Shen M, Du Y. Risk factors for non-syndromic oral clefts: a matched case-control study in Hubei Province, China. Oral Dis. 2015 Jan;21(1):31-7. doi: 10.1111/odi.12200. Epub 2013 Nov 19. PMID 24147616
- [Background] Shilpa G, Gokhale N, Mallineni SK, Nuvvula S. Prevalence of dental anomalies in deciduous dentition and its association with succedaneous dentition: A cross-sectional study of 4180 South Indian children. J Indian Soc Pedod Prev Dent. 2017 Jan-Mar;35(1):56-62. doi: 10.4103/0970-4388.199228. PMID 28139484
- [Background] 4. Tamburini, A. B. F., Rodrigues, Y. H. P., Martelli, D. R. B., de Barros, L. M., de Andrade, R. S., Machado, R. A., Coletta, R. della, Martelli-Júnior, H., & Flório, F. M. (2020). Dental anomalies in the deciduous dentition of non-syndromic oral clefts patients. Revista Brasileira de Saude Materno Infantil, 20(1), 257-263. https://doi.org/10.1590/1806-93042020000100014
- [Background] Tannure PN, Oliveira CA, Maia LC, Vieira AR, Granjeiro JM, Costa Mde C. Prevalence of dental anomalies in nonsyndromic individuals with cleft lip and palate: a systematic review and meta-analysis. Cleft Palate Craniofac J. 2012 Mar;49(2):194-200. doi: 10.1597/10-043. Epub 2011 Jul 8. PMID 21740173